CLINICAL TRIAL: NCT05577208
Title: Cardiac Sympathetic Neuromodulation by Renal Denervation in Hypertrophic Cardiomyopathy (SNYPER Pilot Study)
Brief Title: Renal Denervation in Hypertrophic Cardiomyopathy
Acronym: SNYPER-PS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Adolfo Fontenla (Other)
Responsible Party: Sponsor-Investigator, Adolfo Fontenla, Principal Investigator, Hospital Universitario 12 de Octubre
Organization: Hospital Universitario 12 de Octubre (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNYPER-PS
Record Dates: First submitted 2022-10-06; First posted 2022-10-13 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: renal denervation
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- renal denervation (Experimental): Renal denervation shall be performed by echo-guided catheterization of the femoral artery, and subsequent cannulation of the renal arteries with a guide catheter. A renal denervation catheter shall be advanced through the guide catheter to the distal portion of the artery. The procedures shall be aimed to deliver as many radiofrequency applications as possible, 0.5 cm apart, intended duration of 60 sec, to all four quadrants of the renal arteries and main branch vessels with > 3 mm diameter.
  Interventions: Device: "Symplicity Spyral" multi-electrode renal denervation catheter and "Symplicity G3" generator (Renal Denervation System)

INTERVENTIONS:
Device: "Symplicity Spyral" multi-electrode renal denervation catheter and "Symplicity G3" generator (Renal Denervation System) — Minimally invasive percutaneous interventional therapy aimed to modulate the sympathetic nervous system through endovascular ablation of both renal arteries

SUMMARY:
Hypertrophic cardiomyopathy (HCM) is the most common inherited monogenic heart disease. There is an abnormal increase in myocardial mass in this disorder that leads to a state of cardiac sympathetic hypertonia, which is involved in disease progression, development of arrhythmias and heart failure. Cardiac sympathetic hyperactivity may constitute a new therapeutic target in HCM patients who persist symptomatic despite conventional treatment. The hypothesis of this project is that renal denervation (a minimally invasive percutaneous interventional therapy with proven efficacy in resistant arterial hypertension) reduces cardiac sympathetic activity in HCM. The SNYPER pilot study is a non-randomized clinical trial with medical devices (proof of concept), in which a renal denervation procedure will be performed in 20 patients with genetically confirmed sarcomeric HCM, severe left ventricular hypertrophy and persistent symptoms. The impact of denervation in reducing the 123I-meta iodo benzyl guanidine (MIBG) washout rate quantified by isotopic tracing (planar imaging and SPECT) at 6 months is established as a primary efficacy objective, and the proportion of renal denervation-related complications as a safety objective. The most relevant secondary endpoints are the outcomes of renal denervation on left ventricular mass (echocardiogram), diastolic function, maximum oxygen consumption (ergospirometer), ventricular arrhythmia burden (Holter), blood pressure (ABPM), N-terminal (NT) Pro Brain Natriuretic Peptide (BNP) and quality of life (KCCQ questionnaire). The results of this study may open the development of a new, technically simple and easily accessible therapeutic line for the treatment of HCM.

DETAILED DESCRIPTION:
According to current literature, approximately two-thirds of patients with HCM have persistent symptoms despite conventional treatment. For this reason, novel nonpharmacological therapies such as cardiac resynchronization, endocardial catheter ablation of the interventricular septum or needle-based septal ablation have been proposed, however, none of them having been generalized up to date. Besides, these novel therapies cannot be applied in non-obstructive HCM. The abnormal activation of the sympathetic system represents a relevant mechanism in he pathophysiology of HCM, since it may have implications in the progression and prognosis of the disease. The modulation of the cardiac sympathetic tone by renal denervation could be developed as a new therapeutic target for patients with persistent symptoms despite conventional treatment.

The SNYPER pilot study is a prospective, single-center, single-arm, pilot study, evaluating renal denervation in patients with sarcomeric HCM and persistent symptoms despite optimal therapy, over a follow-up period of 6 months. It represents a proof of concept that will quantify the degree in which renal denervation modulates cardiac sympathetic activity in HCM, thus opening a new research line: a non-pharmacological, minimally invasive and safe treatment with potential positive impact on health and well-being of patients with HCM.

This is a non-commercial, investigator-driven clinical study funded through a public competitive call by Health Institute Carlos III, Spanish Ministry of Economy (PI21/00480).

The study is coordinated by the main investigator from "University Hospital 12 de Octubre" in Madrid. Several responsibilities are delegated to the Clinical Research Unit ("University Hospital 12 de Octubre", Madrid, Spain).

The study was planned according to the Good Clinical Practices. SNYPER Pilot Study has been approved by the Ethics Committee and Spanish Health Authorities. All participating patients must give written informed consent before any study procedure occur.

ELIGIBILITY:
Inclusion Criteria:

1. Sarcomeric HCM (absence of metabolic, syndromic or neurological diseases with increased left ventricular thickness) confirmed by genetic study (pathogenic or probably pathogenic variant identified in a sarcomeric gene).
2. NYHA Class II-IV despite optimal therapy for the last 30 days.
3. Left ventricular septum > 16 mm.
4. Age between 18 and 80 years.
5. Not candidate to septal reduction therapy or valve surgery.

Exclusion Criteria:

1. Non sarcomeric causes of increased left ventricular thickness.
2. Left ventricular systolic disfunction (EF < 50%) or dilatation (indexed left ventricular end diastolic volume [LVEDV] > 75 ml/m2 for men and > 62 ml/m2 for women).
3. Blood pressure < 100/50 mmHg.
4. Severe functional impairment due to concomitant diseases.
5. Renal glomerular filtration < 30 ml/min/m2 (Cockcroft-Gault´s formula).
6. Hospitalization for heart failure, stroke or acute coronary syndrome (ACS) in the last 30 days.
7. Heart failure requiring inotropic drugs or intravenous diuretics over the last 30 days, or in the waiting list for heart transplantation.
8. Unfavorable renal artery anatomy (significant stenosis, diameter < 2mm, length < 4mm)
9. Women on pregnancy, lactation or fertile age without contraception.
10. Parkinson´s disease or Lewy body dementia.
11. Life expectancy less than one year
12. Unwilling to sign informed consent or to undergo study procedure and visits.
13. Participation in other clinical trial over the last 30 days.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-11-26 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiac sympathetic nerve activity (123I-MIBG washout rate) | 6 months
  123I-MIBG washout rate measured by scintigraphy

SECONDARY OUTCOMES:
Functional status | 6 months
  New York Heart Association (NYHA) class. From I to IV (higher scores mean a worse outcome)
Left ventricular mass | 6 months
  Left ventricular mass assessed by echocardiography (Devereux´s formula, septal and posterior wall thickness)
Diastolic function | 6 months
  E / A ratio, deceleration time, E' septal and lateral velocity, E/E´ septal ratio, propagation velocity assessed by echocardiography
Subaortic gradient (left ventricular outflow tract obstruction [LVOT]) | 6 months
  Baseline peak LVOT gradient, peak LVOT gradient during Valsalva in millimeters of mercury
Number of ventricular tachycardia episodes | 6 months
  Non-sustained ventricular tachycardias episodes recorded by a cardiac electronic implantable device (pacemaker or defibrillator, if previously implanted)
Heart rate variability | 6 months
  Number of atrial premature complexes and number of non-sustained atrial tachycardias recorded by 24-hour Holter
Maximum oxygen consumption | 6 months
  Maximum oxygen consumption assessed by ergospirometer
Blood pressure | 6 months
  Mean, daily and nocturnal systolic and diastolic blood pressure assessed by 24-hour ambulatory monitoring of blood pressure (AMBP)
NT-Pro-BNP | 6 months
  Serum NT-Pro-BNP levels
Kansas City Cardiomyopathy Questionnaire (KCCQ) score | 6 months
  Self-administered health-related quality of life questionnaire composed by 23 items, which provides a score range from 0 to 100.

CONTACTS AND LOCATIONS:
Overall Officials: Adolfo Fontenla, MD, PhD, Study Chair — Hospital Universitario 12 de Octubre; Adolfo Fontenla, MD, PhD, Principal Investigator — Hospital Universitario 12 de Octubre
Locations (1):
- Hospital Universitario 12 de Octubre, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
10 milliliters (mL) of total blood, 5mL of serum and 10mL of blood with a commercial formula for RNA preservation shall be collected and stored for future proteomic and genetic analysis.
Supporting Information: Analytic Code
Time Frame: not defined
Access Criteria: not defined

REFERENCES:
- [Background] Lefroy DC, de Silva R, Choudhury L, Uren NG, Crake T, Rhodes CG, Lammertsma AA, Boyd H, Patsalos PN, Nihoyannopoulos P, et al. Diffuse reduction of myocardial beta-adrenoceptors in hypertrophic cardiomyopathy: a study with positron emission tomography. J Am Coll Cardiol. 1993 Nov 15;22(6):1653-60. doi: 10.1016/0735-1097(93)90591-n. PMID 8227834
- [Background] Schafers M, Dutka D, Rhodes CG, Lammertsma AA, Hermansen F, Schober O, Camici PG. Myocardial presynaptic and postsynaptic autonomic dysfunction in hypertrophic cardiomyopathy. Circ Res. 1998 Jan 9-23;82(1):57-62. doi: 10.1161/01.res.82.1.57. PMID 9440705
- [Background] Li ST, Tack CJ, Fananapazir L, Goldstein DS. Myocardial perfusion and sympathetic innervation in patients with hypertrophic cardiomyopathy. J Am Coll Cardiol. 2000 Jun;35(7):1867-73. doi: 10.1016/s0735-1097(00)00626-4. PMID 10841237
- [Background] Taki J, Nakajima K, Bunko H, Simizu M, Muramori A, Hisada K. Whole-body distribution of iodine 123 metaiodobenzylguanidine in hypertrophic cardiomyopathy: significance of its washout from the heart. Eur J Nucl Med. 1990;17(5):264-8. doi: 10.1007/BF00812368. PMID 2128050
- [Background] Pace L, Betocchi S, Losi MA, Della Morte AM, Ciampi Q, Nugnez R, Chiariello M, Salvatore M. Sympathetic nervous function in patients with hypertrophic cardiomyopathy assessed by [123I]-MIBG: relationship with left ventricular perfusion and function. Q J Nucl Med Mol Imaging. 2004 Mar;48(1):20-5. PMID 15195000
- [Background] Rapacciuolo A, Esposito G, Caron K, Mao L, Thomas SA, Rockman HA. Important role of endogenous norepinephrine and epinephrine in the development of in vivo pressure-overload cardiac hypertrophy. J Am Coll Cardiol. 2001 Sep;38(3):876-82. doi: 10.1016/s0735-1097(01)01433-4. PMID 11527648
- [Background] Shimizu M, Ino H, Okeie K, Yamaguchi M, Hayashi K, Nagata M, Itoh H, Iwaki T, Oe K, Konno T, Mabuchi H. Septal wall thinning and systolic dysfunction in patients with hypertrophic cardiomyopathy caused by a cardiac troponin I gene mutation. Am Heart J. 2002 Apr;143(4):690-5. doi: 10.1067/mhj.2002.120291. PMID 11923807
- [Background] Terai H, Shimizu M, Ino H, Yamaguchi M, Uchiyama K, Oe K, Nakajima K, Taki J, Kawano M, Mabuchi H. Changes in cardiac sympathetic nerve innervation and activity in pathophysiologic transition from typical to end-stage hypertrophic cardiomyopathy. J Nucl Med. 2003 Oct;44(10):1612-7. PMID 14530475
- [Background] Hiasa G, Hamada M, Saeki H, Ogimoto A, Ohtsuka T, Hara Y, Shigematsu Y. Cardiac sympathetic nerve activity can detect congestive heart failure sensitively in patients with hypertrophic cardiomyopathy. Chest. 2004 Sep;126(3):679-86. doi: 10.1378/chest.126.3.679. PMID 15364742
- [Background] Terai H, Shimizu M, Ino H, Yamaguchi M, Hayashi K, Sakata K, Kiyama M, Hayashi T, Inoue M, Taki J, Mabuchi H. Cardiac sympathetic nerve activity in patients with hypertrophic cardiomyopathy with malignant ventricular tachyarrhythmias. J Nucl Cardiol. 2003 May-Jun;10(3):304-10. doi: 10.1016/s1071-3581(03)00362-3. PMID 12794630
- [Background] Bhatt DL, Kandzari DE, O'Neill WW, D'Agostino R, Flack JM, Katzen BT, Leon MB, Liu M, Mauri L, Negoita M, Cohen SA, Oparil S, Rocha-Singh K, Townsend RR, Bakris GL; SYMPLICITY HTN-3 Investigators. A controlled trial of renal denervation for resistant hypertension. N Engl J Med. 2014 Apr 10;370(15):1393-401. doi: 10.1056/NEJMoa1402670. Epub 2014 Mar 29. PMID 24678939
- [Background] Kandzari DE, Bohm M, Mahfoud F, Townsend RR, Weber MA, Pocock S, Tsioufis K, Tousoulis D, Choi JW, East C, Brar S, Cohen SA, Fahy M, Pilcher G, Kario K; SPYRAL HTN-ON MED Trial Investigators. Effect of renal denervation on blood pressure in the presence of antihypertensive drugs: 6-month efficacy and safety results from the SPYRAL HTN-ON MED proof-of-concept randomised trial. Lancet. 2018 Jun 9;391(10137):2346-2355. doi: 10.1016/S0140-6736(18)30951-6. Epub 2018 May 23. PMID 29803589
- [Background] Bohm M, Kario K, Kandzari DE, Mahfoud F, Weber MA, Schmieder RE, Tsioufis K, Pocock S, Konstantinidis D, Choi JW, East C, Lee DP, Ma A, Ewen S, Cohen DL, Wilensky R, Devireddy CM, Lea J, Schmid A, Weil J, Agdirlioglu T, Reedus D, Jefferson BK, Reyes D, D'Souza R, Sharp ASP, Sharif F, Fahy M, DeBruin V, Cohen SA, Brar S, Townsend RR; SPYRAL HTN-OFF MED Pivotal Investigators. Efficacy of catheter-based renal denervation in the absence of antihypertensive medications (SPYRAL HTN-OFF MED Pivotal): a multicentre, randomised, sham-controlled trial. Lancet. 2020 May 2;395(10234):1444-1451. doi: 10.1016/S0140-6736(20)30554-7. Epub 2020 Mar 29. PMID 32234534
- [Background] Fontenla A, Garcia-Donaire JA, Hernandez F, Segura J, Salgado R, Cerezo C, Ruilope LM, Arribas F. Management of resistant hypertension in a multidisciplinary unit of renal denervation: protocol and results. Rev Esp Cardiol (Engl Ed). 2013 May;66(5):364-70. doi: 10.1016/j.rec.2012.09.006. Epub 2012 Dec 11. PMID 24775818
- [Background] Rodriguez-Leor O, Segura J, Garcia Donaire JA, Gutierrez-Ibanes E, Oliveras A, Mediavilla JD, Serrador A, Prado JC, Nunez-Gil I, Diez-Delhoyo F, Clara Velasco A, Jaen Aguila F, Amat-Santos I, Bayes-Genis A, Troya Saborido MI. Renal denervation for the treatment of resistant hypertension in Spain. The Flex-Spyral Registry. Rev Esp Cardiol (Engl Ed). 2020 Aug;73(8):615-622. doi: 10.1016/j.rec.2019.08.001. Epub 2019 Sep 24. English, Spanish. PMID 31561981
- [Background] Donazzan L, Mahfoud F, Ewen S, Ukena C, Cremers B, Kirsch CM, Hellwig D, Eweiwi T, Ezziddin S, Esler M, Bohm M. Effects of catheter-based renal denervation on cardiac sympathetic activity and innervation in patients with resistant hypertension. Clin Res Cardiol. 2016 Apr;105(4):364-71. doi: 10.1007/s00392-015-0930-4. Epub 2015 Oct 22. PMID 26493305
- [Background] Armaganijan LV, Staico R, Moreira DA, Lopes RD, Medeiros PT, Habib R, Melo Neto J, Katz M, Armaganijan D, Sousa AG, Mahfoud F, Abizaid A. 6-Month Outcomes in Patients With Implantable Cardioverter-Defibrillators Undergoing Renal Sympathetic Denervation for the Treatment of Refractory Ventricular Arrhythmias. JACC Cardiovasc Interv. 2015 Jun;8(7):984-90. doi: 10.1016/j.jcin.2015.03.012. PMID 26088516
- [Background] Steinberg JS, Shabanov V, Ponomarev D, Losik D, Ivanickiy E, Kropotkin E, Polyakov K, Ptaszynski P, Keweloh B, Yao CJ, Pokushalov EA, Romanov AB. Effect of Renal Denervation and Catheter Ablation vs Catheter Ablation Alone on Atrial Fibrillation Recurrence Among Patients With Paroxysmal Atrial Fibrillation and Hypertension: The ERADICATE-AF Randomized Clinical Trial. JAMA. 2020 Jan 21;323(3):248-255. doi: 10.1001/jama.2019.21187. PMID 31961420
- [Background] Chen W, Ling Z, Xu Y, Liu Z, Su L, Du H, Xiao P, Lan X, Shan Q, Yin Y. Preliminary effects of renal denervation with saline irrigated catheter on cardiac systolic function in patients with heart failure: A Prospective, Randomized, Controlled, Pilot Study. Catheter Cardiovasc Interv. 2017 Mar 1;89(4):E153-E161. doi: 10.1002/ccd.26475. Epub 2016 May 3. PMID 27143319
- [Background] Mahfoud F, Urban D, Teller D, Linz D, Stawowy P, Hassel JH, Fries P, Dreysse S, Wellnhofer E, Schneider G, Buecker A, Schneeweis C, Doltra A, Schlaich MP, Esler MD, Fleck E, Bohm M, Kelle S. Effect of renal denervation on left ventricular mass and function in patients with resistant hypertension: data from a multi-centre cardiovascular magnetic resonance imaging trial. Eur Heart J. 2014 Sep 1;35(33):2224-31b. doi: 10.1093/eurheartj/ehu093. Epub 2014 Mar 6. PMID 24603307
- [Background] Schirmer SH, Sayed MM, Reil JC, Lavall D, Ukena C, Linz D, Mahfoud F, Bohm M. Atrial Remodeling Following Catheter-Based Renal Denervation Occurs in a Blood Pressure- and Heart Rate-Independent Manner. JACC Cardiovasc Interv. 2015 Jun;8(7):972-80. doi: 10.1016/j.jcin.2015.02.014. Epub 2015 May 20. PMID 26003031
- [Background] Cardim N, Brito D, Rocha Lopes L, Freitas A, Araujo C, Belo A, Goncalves L, Mimoso J, Olivotto I, Elliott P, Madeira H; participating centres. The Portuguese Registry of Hypertrophic Cardiomyopathy: Overall results. Rev Port Cardiol (Engl Ed). 2018 Jan;37(1):1-10. doi: 10.1016/j.repc.2017.08.005. Epub 2018 Jan 19. English, Portuguese. PMID 29358015
- [Background] Wenning C, Lange PS, Schulke C, Vrachimis A, Monnig G, Schober O, Eckardt L, Schafers M. Pulmonary vein isolation in patients with paroxysmal atrial fibrillation is associated with regional cardiac sympathetic denervation. EJNMMI Res. 2013 Dec 21;3(1):81. doi: 10.1186/2191-219X-3-81. PMID 24360192